CLINICAL TRIAL: NCT05207033
Title: Young Adults' Responses to E-Cigarette Advertisement Features and the Effect of Restricting Features on Tobacco Use - Phase 2
Brief Title: Responses to Regulated E-Cigarette Advertisements
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Elise Stevens, Assistant Professor, University of Massachusetts, Worcester
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: H00022520; 4R00DA046563-04 (NIH)
Record Dates: First submitted 2021-12-15; First posted 2022-01-26 (Actual); Results first posted 2025-05-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Tobacco Use
MeSH Terms: conditions — Tobacco Use

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Unregulated ad condition (Active Comparator): This arm will include exposure to unregulated e-cigarette ads or ads as they appear in modern media.
  Interventions: Other: Unregulated ad condition
- Regulated ad condition (Experimental): This arm will include exposure to regulated e-cigarette ads or ads where we have taken out the appealing features.
  Interventions: Other: Regulated ad condition

INTERVENTIONS:
Other: Regulated ad condition — This intervention will determine if restriction of appealing features in e-cigarette ads deter young adults from trying the product.
  Arms: Regulated ad condition
Other: Unregulated ad condition — This intervention will determine if unrestricted appealing features in e-cigarette ads deter young adults from trying the product.
  Arms: Unregulated ad condition

SUMMARY:
While conventional cigarette use continues to decline among youth and young adults, e-cigarette (EC) use is on the rise. Specifically, the investigators will conduct a randomized control trial (RCT) where young adults are randomized to one of two conditions: 1) a regulated ad environment, with high impact EC ad features removed or 2) an unregulated ad environment, with high impact EC ad features left intact. Participants will view EC ads embedded in an online magazine 24 times over the course of 6 months. EC experimentation and sustained use will be the primary outcome of interest.

DETAILED DESCRIPTION:
While conventional cigarette use continues to decline among youth and young adults, e-cigarette (EC) use is on the rise. The use of ECs during young adulthood, particularly 18 years of age, is especially alarming because it is not only a critical period in development but also a time when tobacco use is established. Additionally, the tobacco industry targets individuals of this age with the hope that they will one day progress to using combustible cigarettes. Advertising may be one of the reasons leading young people to use ECs, and the Food and Drug Administration (FDA) now has the authority to regulate EC advertisement features. The goal of the proposed study is to determine which EC ad features most strongly influence young adults' attitudes, susceptibility, and intentions to use ECs, and determine if the restriction of these ad features influences EC attitudes, experimentation, and sustained use. The investigators will experimentally estimate the causal effect of restricting high impact EC ad features on tobacco use behavior. Specifically, the investigators will conduct a randomized control trial (RCT) where young adults are randomized to one of two conditions: 1) a regulated ad environment, with high impact EC ad features removed or 2) an unregulated ad environment, with high impact EC ad features left intact. Participants will view EC ads embedded in an online magazine 24 times over the course of 6 months. EC experimentation and sustained use will be the primary outcome of interest. We will also examine how sensation seeking, impulsivity, and sleep health impact EC use. Findings from this study will provide public health officials important and urgently needed information as to what advertising features are contributing to the sharp rise in the use of ECs among young adults, and if restrictions reduce the use of ECs among young adults.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 26 years old,
* fluent in English (earn a score of at least 4 on the Rapid Estimate of Adult Literacy in Medicine)
* biochemically confirmed abstinence of alcohol (BrAC=.00) and combusted tobacco or marijuana exhaled carbon monoxide (eCO<6 parts per million) at time of visit,
* reporting never trying an e-cigarette, not even a puff OR reporting tried and e-cigarette in the past but not in the past 30 days. Susceptibility to EC use, will be determined using the Susceptibility to Use Tobacco Products questionnaire, with only those identifying anything besides "no curiosity/interest" to all three susceptibility questions as susceptible users.

Exclusion Criteria:

* Out of age range 18-26 years
* Use of an e-cigarette in past 30 days
* Pregnant women

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 195 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-06-04 (Actual); Study Completion 2024-07-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UMass Chan Medical School Stevens Lab, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Enrollment was N=195, however, prior to assignment, 9 participants stopped responding to communications from study staff including the initial survey, and thus were never assigned to a arm/group.
Period: Overall Study
Arm/Group | Unregulated ad Condition | Regulated ad Condition
Started | 94 | 92
Completed | 88 | 84
Not Completed | 6 | 8

BASELINE CHARACTERISTICS:
Population: Participants were included in the analysis if they had at least baseline and 6-month data.
Groups:
- Total: Total of all reporting groups
Arm/Group | Unregulated ad Condition | Regulated ad Condition | Total
Number analyzed (Participants) | 88 | 84 | 172
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 88 | 84 | 172
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.13 (2.32) | 22.88 (2.54) | 22.5 (2.46)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  female | 67 | 69 | 136
  male | 16 | 13 | 29
  other | 5 | 2 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 7 | 18 | 25
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 8 | 9
  White | 57 | 44 | 101
  More than one race | 7 | 10 | 17
  Unknown or Not Reported | 16 | 4 | 20
Region of Enrollment [Number; unit: participants]
  United States | 88 | 84 | 171

OUTCOME MEASURES:

1. Primary Outcome: Tobacco Use at 1 Month
Description: Use of any tobacco products
Time Frame: 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | Unregulated ad Condition | Regulated ad Condition
Number analyzed (Participants) | 87 | 84
Participants | 5 | 5

2. Primary Outcome: Tobacco Use at 3 Months
Description: Use of any tobacco products
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Unregulated ad Condition | Regulated ad Condition
Number analyzed (Participants) | 87 | 84
Participants | 3 | 2

3. Primary Outcome: Tobacco Use at 6 Months
Description: Use of any tobacco products
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Unregulated ad Condition | Regulated ad Condition
Number analyzed (Participants) | 87 | 84
Participants | 1 | 2

4. Primary Outcome: Perceived Severity of Using E-Cigarettes at 1 Month
Description: Perceived severity of using e-cigarettes, a subconstruct of the Health Belief Model was assessed by participants' perceived significance, severity, and seriousness of health threats from e-cigarette use. The measure is as follows in its exact and unabbreviated form:
  Please rate the following statements on a scale from 1 (strongly disagree) to 5 (strongly agree).
  I believe that the health threat of using e-cigarettes is severe. I believe that the health threat of using e-cigarettes is serious. I believe that the health threat of using e-cigarettes is significant.
  To determine score, the average is taken of the items. Minimum Score = 1; Maximum Score = 5 Higher scores indicate greater perceived severity of e-cigarette use. Lower scores indicate lesser perceived severity of e-cigarette use.
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Unregulated ad Condition | Regulated ad Condition
Number analyzed (Participants) | 87 | 84
units on a scale | 4.41 (.66) | 4.46 (.61)

5. Primary Outcome: Perceived Severity of Using E-Cigarettes at 3 Months
Description: as for outcome 4
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Unregulated ad Condition | Regulated ad Condition
Number analyzed (Participants) | 87 | 84
units on a scale | 4.41 (.67) | 4.36 (.71)

6. Primary Outcome: Perceived Severity of Using E-Cigarettes at 6 Months
Description: as for outcome 4
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Unregulated ad Condition | Regulated ad Condition
Number analyzed (Participants) | 87 | 84
units on a scale | 4.48 (.63) | 4.48 (.59)

7. Primary Outcome: Motivation to Avoid E-Cigarettes at 1 Month
Description: Motivation to avoid e-cigarettes was assessed by participants' self-reported importance, confidence, readiness, and commitment to avoid e-cigarette use in the future. These items reflect constructs from behavior change theories such as the Transtheoretical Model, which emphasizes individual readiness and self-efficacy as key predictors of behavioral intention and action. The measure is as follows in its exact and unabbreviated form:
  Please rate the following statements on a scale from 0 to 10. 0 = Not at all 10 = Very
  How important is it to avoid e-cigarettes in the future?
  How confident are you in avoiding e-cigarettes in the future?
  How ready are you to avoid e-cigarettes in the future?
  How committed are you to avoid e-cigarettes in the future?
  To determine score, the average is taken across the four items. Minimum Score = 0; Maximum Score = 10 Higher scores indicate greater motivation to avoid e-cigarette use. Lower scores indicate lesser motivation.
Time Frame: 1 Month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Unregulated ad Condition | Regulated ad Condition
Number analyzed (Participants) | 87 | 84
score on a scale | 7.66 (2.03) | 8.05 (1.89)

8. Primary Outcome: Motivation to Avoid E-Cigarettes at 3 Months
Description: as for outcome 7
Time Frame: 3 Months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Unregulated ad Condition | Regulated ad Condition
Number analyzed (Participants) | 87 | 84
score on a scale | 7.74 (2.13) | 8.02 (1.87)

9. Primary Outcome: Motivation to Avoid E-Cigarettes at 6 Months
Description: as for outcome 7
Time Frame: 6 Months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Unregulated ad Condition | Regulated ad Condition
Number analyzed (Participants) | 87 | 84
score on a scale | 7.87 (2.08) | 8.00 (1.87)

10. Primary Outcome: Behavioral Intentions at 1 Month
Description: Behavioral intentions to use e-cigarettes were assessed using participants' self-reported interest and willingness to engage in future e-cigarette use. This construct is grounded in the Theory of Planned Behavior, which identifies behavioral intention as the most immediate and reliable predictor of future behavior. The measure is as follows in its exact and unabbreviated form:
  How interested are you in trying e-cigarettes?
  How willing are you to try e-cigarettes?
  How willing would you be to purchase an e-cigarette?
  How willing would you be to try an e-cigarette if a friend offered you one?
  Responses were rated on a scale from 1 (not at all) to 5 (very). To determine score, the average is taken across the four items. Minimum Score = 1; Maximum Score = 5 Higher scores indicate stronger behavioral intentions to use e-cigarettes. Lower scores indicate weaker intentions.
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Unregulated ad Condition | Regulated ad Condition
Number analyzed (Participants) | 87 | 84
score on a scale | 3.23 (.76) | 3.32 (.76)

11. Primary Outcome: Behavioral Intentions at 3 Months
Description: as for outcome 10
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Unregulated ad Condition | Regulated ad Condition
Number analyzed (Participants) | 87 | 84
score on a scale | 3.19 (.83) | 3.37 (.80)

12. Primary Outcome: Behavioral Intentions at 6 Months
Description: as for outcome 10
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Unregulated ad Condition | Regulated ad Condition
Number analyzed (Participants) | 87 | 84
score on a scale | 3.24 (.75) | 3.20 (.88)

13. Primary Outcome: Number of Participants With Biochemical Verification of Tobacco Use at 1 Month
Description: Biochemical confirmation of tobacco use was conducted using the Alere iScreen Oral Fluid Device (OFD), a point-of-care saliva test that detects cotinine, a primary metabolite of nicotine, indicating tobacco or nicotine product use within the past ~3 days. The count reflects participants who tested positive for cotinine, providing biochemical evidence of recent tobacco or nicotine exposure.
Time Frame: 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | Unregulated ad Condition | Regulated ad Condition
Number analyzed (Participants) | 87 | 84
Participants | 0 | 1

14. Primary Outcome: Number of Participants With Biochemical Verification of Tobacco Use at 3 Months
Description: as for outcome 13
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Unregulated ad Condition | Regulated ad Condition
Number analyzed (Participants) | 87 | 84
Participants | 1 | 2

15. Primary Outcome: Number of Participants With Biochemical Verification of Tobacco Use at 6 Months
Description: as for outcome 13
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Unregulated ad Condition | Regulated ad Condition
Number analyzed (Participants) | 87 | 84
Participants | 0 | 3

ADVERSE EVENTS:
Time Frame: Adverse events were collected over the course of 6 months.
Arm/Group | Unregulated ad Condition | Regulated ad Condition
All-Cause Mortality (participants affected / at risk) | 0/94 | 0/92
Serious Adverse Events (participants affected / at risk) | 0/94 | 0/92
Other Adverse Events (participants affected / at risk) | 0/94 | 0/92

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-04-03): https://cdn.clinicaltrials.gov/large-docs/33/NCT05207033/Prot_SAP_000.pdf